CLINICAL TRIAL: NCT05094895
Title: Radiofrequency Energy Delivery to the Gastro-esophageal Junction (Stretta®) in Gastro-esophageal Reflux Disease After Sleeve Gastrectomy
Brief Title: Stretta Treatment in GERD After SG
Acronym: Stretta
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Timshel BV (Unknown)
Responsible Party: Principal Investigator, Prof Dr Jan Tack, Prof. Dr., Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S64212
Record Dates: First submitted 2021-10-20; First posted 2021-10-26 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Stretta Device
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Patients will receive the Stretta treatment or the Sham treatment. Patients assigned to the Sham treatment condition, will have an open label period and are able to receive the Stretta treatment as wel.
Who Masked: Participant, Care Provider
Masking Description: In the first period are the patients and investigators blinded. Afterwards there is an open label period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Stretta Treatment (Active Comparator): Patients will receive the Stretta treatment
  Interventions: Procedure: Stretta
- Sham treatment (Sham Comparator): Patients will receive the sham treatment
  Interventions: Procedure: Sham

INTERVENTIONS:
Procedure: Stretta — Radiofrequency energy delivered to the gastro-esophageal junction
  Arms: Stretta Treatment
Procedure: Sham — Patients that have the sham condition will have a procedure using a 24Fr Savary bougie dilator over the guidewire, with the same sedation.
  Arms: Sham treatment

SUMMARY:
To evaluate the effect and explore the mechanism of action behind the potential effect of Stretta® on GERD after SG.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD), i.e. the occurrence of troublesome symptoms or lesions as a consequence of retrograde flow of gastric contents into the esophagus, is one of the most prevalent gastrointestinal disorders. Obesity, defined by a body mass index (BMI) of ≥ 30 kg/m2, is an increasingly important problem in the Western world and a well-known risk factor for GERD related symptoms and esophagitis. Possible underlying mechanisms include an increased gastroesophageal pressure gradient, upward positional shift of the lower esophageal sphincter (LES) and increased occurrence of transient LES relaxations (TLESRs) after a meal.

Bariatric surgery has emerged as a highly effective treatment for obesity and its associated metabolic complications. Roux-en-Y gastric bypass and sleeve gastrectomy (SG) currently account for the majority of the procedures. Several studies have reported improvement of GERD after gastric bypass and SG, probably through a combination of reduction of the acid-producing gastric mucosa and weight loss. However, in up to 34% of patients who underwent SG, de novo GERD or worsening of pre-existent GERD becomes evident, which established baseline GERD symptoms one of the few relative contra-indications for SG in many centers. Several post-operative alterations have been hypothesized to explain the increased incidence of GERD after SG: increased incidence of hiatal hernia due to the sleeve formation, dissection of the phreno-esophageal ligament, intrathoracic sleeve migration, increased intragastric pressure due to decreased gastric compliance and disruption of the competency of the esophagogastric junction (EGJ).

Despite the fact that the majority of patients will respond to proton pump inhibitor (PPI) therapy, a significant proportion of patients continue to experience regurgitation and/or heartburn despite acid suppression although treatment outcome data are largely missing in the literature. These patients with refractory GERD symptoms after SG pose a challenge to surgeons and gastroenterologists since the postoperative anatomy does not allow classic fundoplication procedures.

Stretta® (Mederi RF LLC, Houston TX, USA) is an endoscopic anti-reflux procedure using the delivery of radiofrequency energy to the LES. Stretta® is supported by the Society of American Gastrointestinal Endoscopic Surgeons (SAGES, ASGE and NICE) for the treatment of GERD in selected patients and is long-term cost-effective. Several controlled studies and a meta-analysis have reported improved symptoms after Stretta® although the effect on esophageal acid exposure time is inconsistent. Stretta® decreases the compliance of the EGJ without inducing fibrosis since the effect was reversed by administration of a nitric oxide donor and decreased sensitivity to distal acid perfusion. However, studies evaluating the symptomatic benefit of Stretta® in patients after SG are lacking, which is the primary goal of our study (primary endpoint). With the secondary endpoints, the effect of Stretta® will also be investigated on various aspects, which will provide an insight in the mechanism of action behind the potential effect of the intervention.

ELIGIBILITY:
Inclusion Criteria:

1. 18 to 65 years old;
2. History of typical GERD symptoms (heartburn or regurgitation) during PPI treatment, at least 3 times per week for 12 weeks ('refractory GERD') or unwillingness to take/continue PPIs. The symptoms can be de novo (onset after sleeve gastrectomy) or pre-existing (as documented by medication use, findings during endoscopy or medical history);
3. In case of refractory GERD symptoms during PPI treatment the following criteria need to be fulfilled: Pathological catheter-based 24h pH-MII monitoring off-PPI (>6% of total time pH<4 and/or number of reflux episodes >80 (irrespective of acidity) or positive symptom association probability (SAP) for typical reflux symptoms) based on the Lyon consensus (23);
4. More than 12 months after sleeve gastrectomy;
5. Willing to take contraceptive measurements.

Exclusion Criteria:

1. Hiatal hernia of >2cm as determined during HRiM (based on Chicago Classification v3.0. (24)) and/or endoscopy or hiatal hernia repair;
2. Esophagitis LA classification grade C or D during gastroscopy off-PPI;
3. Circumferential Barrett's esophagus >1cm (columnar lined esophageal mucosa with intestinal metaplasia) or history of ablation of Barrett's esophagus;
4. Esophageal or fundus varices during gastroscopy;
5. Esophageal strictures during gastroscopy;
6. Abnormalities in sleeve (e.g. sleeve migration) observed during gastroscopy and/or barium test;
7. Known cirrhosis or portal hypertension from other causes;
8. History of surgery to the upper gastrointestinal tract other than sleeve gastrectomy, including redo after previous bariatric surgery;
9. Autoimmune or a connective tissue disorder (scleroderma, dermatomyositis, Calcinosis-Raynaud's-Esophagus Sclerodactily Syndrome (CREST), Sjogren's Syndrome, etc.);
10. Achalasia, EGJ-outflow obstruction, jackhammer esophagus or absent contractility as defined by the 3rd revision of the Chicago classification for primary esophageal motility disorders24 assessed during HRiM with meal (see study protocol (25));
11. Significant cardiopulmonary or other comorbidity precluding safe sedation;
12. Pacemaker or implanted cardiac defibrillator;
13. Coagulopathy or use of anticoagulants;
14. Pregnancy or breastfeeding
15. Unable or unwilling to consent for an invasive procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-29 (Actual); Primary Completion 2024-01-29 (Estimated); Study Completion 2024-01-29 (Estimated)

PRIMARY OUTCOMES:
Symptom severity | ReQuest questionnaire score will be assessed at week -1 after treatment
  Primary efficacy endpoint will be the change in symptom severity assessed by validated reflux questionnaires (ReQuest questionnaire and diaries) at week -1
Symptom severity | ReQuest questionnaire score will be assessed at week 12 after treatment
  Primary efficacy endpoint will be the change in symptom severity assessed by validated reflux questionnaires (ReQuest questionnaire and diaries) at week 12
Symptom severity | ReQuest questionnaire score will be assessed at week 24 after treatment
  Primary efficacy endpoint will be the change in symptom severity assessed by validated reflux questionnaires (ReQuest questionnaire and diaries) at week 24
Symptom severity | ReQuest questionnaire score will be assessed at 1 year after treatment
  Primary efficacy endpoint will be the change in symptom severity assessed by validated reflux questionnaires (ReQuest questionnaire and diaries) 1 year after treatment

SECONDARY OUTCOMES:
Objective reflux parameters | Will be assessed week -1, week 12 and week 24
  change in the objective reflux parameters on 24h pH-impedance (pH-MII) measurement
High Resolution impedance manometry | Will be assessed week -1 and week 24
  Change in HRiM paramters
EGJ distensibility (Endoflip) | Will be assessed week -1 and week 24
  Change in EGJ distensibility
Esophageal sensitivity | Will be assessed week -1 and week 24
  Change in esophageal sensitivity
Esophageal permeability | Will be assessed week -1 and week 24
  Change in esophageal permeability assessed by transepithelial electrical resistance
Microscopic esophagitis (ESOHISTO score) | Will be assessed week -1 and week 24
  Change in esophagitis using esohisto scoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Annelies Geeraerts, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided